CLINICAL TRIAL: NCT07309302
Title: Psychosocial Determinants and Impact of a Synchronous Remote Cognitive Remediation Program on Individuals With Post-Traumatic Stress Disorder.
Brief Title: Psychosocial Factors and Efficacy of Remote Cognitive Remediation for Post-Traumatic Stress Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Responsible Party: Principal Investigator, Pascale Brillon, Ph.D., Principal Investigator, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-5811
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: Cognitive remediation; Social Support; Quality of Life; Online Intervention; Self-Efficacy; Depression; Anxiety; Attention; Verbal Memory; Executive Functions; Life Satisfaction; Post-Traumatic Stress Disorder; Neuropsychological functions
MeSH Terms: conditions — Combat Disorders; Depression; Anxiety Disorders; Personal Satisfaction; Stress Disorders, Post-Traumatic | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation Training (Experimental): Cognitive Remediation Training
  Interventions: Behavioral: Cognitive Remediation Training
- Video Games with Life Quality Support (Placebo Comparator): Video Games with Quality of Life Support
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Cognitive Remediation Training — Cognitive Remediation Training: Eight-week remote program using HAPPYneuron Pro software targeting attention, verbal memory, processing speed, and executive functions.
  Participants attend weekly 75-minute group sessions (maximum six participants) via videoconferencing: 30 minutes of computerized cognitive exercises and 45 minutes of guided discussion on metacognitive strategies and quality-of-life topics. Weekly homework assignments (45 minutes) reinforce skills. Sessions target attention (selective, sustained, divided), verbal memory (encoding, recall, recognition), and executive functions (planning, problem-solving, cognitive flexibility, inhibition).
  Strategy teachings address attention, verbal memory, planning, problem-solving, emotion regulation, meditation, and cognitive flexibility. Quality of life discussions (summarized format) cover sleep, nutrition, physical activity, social support, cultural activities, nature-based activities, relaxation, and substance use behaviors.
  Arms: Cognitive Remediation Training
Other: Control Group — Video Games with Quality of Life Support: Eight-week active control program combining commercial video games with quality of life discussions. Participants will attend weekly 75-minute group sessions via secure videoconferencing (maximum of six participants), consisting of 30 minutes of entertaining computer games from the Poki.com platform (games include Bubbles, Sweet World, Minesweeper, etc.) and 45 minutes of group discussions on healthy lifestyle topics including sleep, nutrition, physical activity, social support, cultural activities, nature-based activities, relaxation, and substance use behaviors. Weekly individual gaming assignments (30 minutes) maintain engagement. Games are selected for entertainment value without proven cognitive benefits. Discussions focus on general wellness and lifestyle factors rather than cognitive strategy development.
  Arms: Video Games with Life Quality Support

SUMMARY:
The goal of this clinical trial is to evaluate whether computer-based brain training can help adults with post-traumatic stress disorder (PTSD). Individuals with PTSD often experience difficulties with memory, attention, concentration, and problem-solving, which can significantly affect their daily lives, work performance, and overall quality of life. These cognitive challenges can hinder trauma recovery and reduce the effectiveness of standard PTSD treatments.

The main questions this study seeks to address are:

Does specialized brain training improve PTSD symptoms compared to regular computer games? Does brain training enhance cognitive functions such as memory, attention, processing speed, and executive functioning? Does brain training improve quality of life and daily functioning? Do participants' self-efficacy and perceived social support influence treatment outcomes?

Researchers will compare two approaches: a specialized cognitive training program (HAPPYneuron Pro) with strategy teachings and quality-of-life discussions, versus engaging computer games with quality-of-life discussions, to determine which is more effective for people with PTSD.

Study Design

Participants will be randomly assigned to one of two groups for an 8-week program:

Cognitive remediation training group: Complete computerized cognitive exercises and strategy teachings specifically designed to strengthen memory, attention, and executive functions, combined with quality-of-life discussions.

Control group: Complete engaging computer games combined with quality-of-life discussions.

Schedule

Both groups will follow the same schedule:

One online session per week, in small and consistent groups of 6 participants. Each 60-minute session consists of 30 minutes of computer activities followed by 45 minutes of group discussion.

One at-home individual homework exercise per week (30 minutes at home).

Total time commitment: 1h45 per week for 8 weeks.

Assessments All participants will complete three comprehensive assessment sessions: before treatment, immediately after the 8-week program, and 3 months later. Assessments include neuropsychological testing and questionnaires on PTSD symptoms, depression, anxiety, quality of life, satisfaction with life, social support, cognitive failures, and self-efficacy.

Significance This research evaluates a new, accessible and remotely deliverable approach for PTSD treatment. Current evidence-based treatments often do not directly target the cognitive impairments experienced by many individuals with PTSD.

Compensation Participants will receive $35 for each completed assessment (maximum $105). Control group participants will gain access to the cognitive remediation training program after completing their participation.

ELIGIBILITY:
Inclusion Criteria

* Age 18 to 45 years
* Able to speak and read French fluently
* Access to a computer with a camera and a secure Internet connection
* Access to a private space for assessment and intervention sessions
* Available for the complete treatment protocol
* Confirmed current PTSD diagnosis using the Structured Clinical Interview for DSM-5 (SCID-5)
* Residing in Canada

Exclusion Criteria

* History of neurological disorders (stroke, intracranial surgery, aneurysm, epilepsy)
* Moderate to severe traumatic brain injury OR hospitalization due to traumatic brain injury
* Mild traumatic brain injury less than 6 months ago with persistent symptoms
* Psychotic disorders
* Alcohol abuse or substance dependence disorders
* Video game addiction
* Hospitalization for major depression or suicide risk within the past 3 months
* Regular use of medications that impact neurocognition, including: benzodiazepines (diazepam, lorazepam, alprazolam, Ativan, Xanax, Rivotril)
* Residence outside Canada

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-08-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Life Scale | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Satisfaction with Life Scale (SWL) is a 5-item self-report questionnaire measuring global life satisfaction. Participants rate their agreement with life satisfaction statements using a 7-point Likert scale (1 = Strongly disagree, 7 = Strongly agree). Total scores range from 5 to 35. Score interpretations: 5-9 (extremely dissatisfied), 10-14 (dissatisfied), 15-19 (slightly dissatisfied), 20 (neutral), 21-25 (slightly satisfied), 26-30 (satisfied), 31-35 (extremely satisfied). Higher scores indicate greater satisfaction with life.
Cognitive Failures Questionnaire | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Cognitive Failures Questionnaire (CFQ) is a 25-item self-report measure assessing the frequency of cognitive lapses and everyday mistakes in memory, attention, and motor function over the past 6 months. Participants rate how often they experience each cognitive failure using a 5-point frequency scale (0 = Never, 1 = Very rarely, 2 = Occasionally, 3 = Quite often, 4 = Very often). Total scores range from 0 to 100, with higher scores indicating more frequent cognitive failures and perceived cognitive dysfunction in daily life. This measure captures subjective cognitive complaints that may not be detected by objective neuropsychological tests.
World Health Organization Quality of Life Scale-Brief | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The World Health Organization Quality of Life Scale-Brief (WHOQOL-BREF) is a 26-item self-report questionnaire assessing four domains of quality of life: Physical Health (7 items, raw score range 7-35), Psychological Health (6 items, raw score range 6-30), Social Relationships (3 items, raw score range 3-15), and Environment (8 items, raw score range 8-40). Two additional items assess overall quality of life and general health. Participants rate items using 5-point Likert scales with varying response options (e.g., 1 = Very poor to 5 = Very good; 1 = Not at all to 5 = Completely). Domain scores are calculated by summing item responses and transforming to a 0-100 scale, where higher scores indicate better quality of life in that domain.
Multidimensional Scale of Perceived Social Support | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item self-report questionnaire measuring perceived social support from three sources: family (4 items), friends (4 items), and significant other (4 items). Participants rate their agreement with each statement over the past 2 weeks using a 7-point Likert scale (1 = Very strongly disagree, 7 = Very strongly agree). The total score ranges from 12 to 84, calculated by summing all item responses. Higher scores indicate greater perceived social support. Score interpretations: 12-36 (low support), 37-60 (moderate support), 61-84 (high support). Subscale scores can also be calculated for each support source (range: 4-28 per subscale).
General Self-Efficacy Scale | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The General Self-Efficacy Scale (GSES) is a 10-item self-report questionnaire measuring general beliefs in one's ability to cope with difficult situations and obstacles. Participants rate how true each statement is for them using a 4-point scale (1 = Not at all true, 2 = Hardly true, 3 = Moderately true, 4 = Exactly true). Total scores range from 10 to 40, calculated by summing all item responses. Higher scores indicate stronger general self-efficacy beliefs. The scale assesses optimistic self-beliefs about coping with demands in various life domains and has been shown to predict adaptation following stressful life events.
Self-Efficacy Scale for Cognitive Remediation Therapy | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Self-Efficacy Scale for Cognitive Remediation Therapy (SE-CRT) is a 7-item self-report questionnaire measuring confidence in successfully completing cognitive remediation exercises. Participants rate their confidence level for each task using a 5-point scale (1 = Not at all confident, 2 = Slightly confident, 3 = Moderately confident, 4 = Very confident, 5
  = Extremely confident). Items assess confidence in maintaining attention, using memory strategies, flexible problem-solving, applying strategies to daily life, time management, performing at average levels, and completing the entire treatment program. Total scores range from 7 to 35, with higher scores indicating greater treatment-specific self-efficacy.
Continuous Performance Test with Rapid Automatized Naming | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Continuous Performance Test with Rapid Automatized Naming (CPT-RAN) is a computerized test of sustained attention and response inhibition from the ExecQC Battery administered via Pavlovia. Participants monitor a continuous stream of rapidly presented stimuli and respond to target stimuli while withholding responses to non-targets. The primary outcome is the d-prime (d') score, a signal detection measure that accounts for both hit rate and false alarm rate, providing a sensitivity index of discriminability between targets and non-targets. Scores typically range from 0 to 5+, with higher values indicating better sustained attention and vigilance. The test also yields reaction time and response consistency measures.
Visual Search Task | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Visual Search Task (VST) is a computerized assessment of visual selective attention, processing speed and visual scanning ability from the ExecQC Battery administered via Pavlovia. Participants search for a target stimulus among distractors in visual arrays of varying complexity (set sizes). The primary outcomes are: (1) mean reaction time in milliseconds for correct target detection (lower = better performance), and (2) accuracy percentage (higher = better performance). The search slope (change in reaction time as set size increases) provides additional information about search efficiency and attentional capacity.
Trail Making Test | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Trail Making Test (TMT) is a computerized version from the ExecQC Battery administered via Pavlovia, measuring processing speed, visual scanning and executive functions. Part A requires connecting numbered circles in ascending order (1-2-3...), assessing processing speed and visual attention. Part B requires alternating between numbers and letters (1-A-2-B-3-C...), assessing cognitive flexibility and set-shifting. Primary outcomes are completion times in seconds for each part (lower = better performance). The difference score (Part B minus Part A) isolates executive function independent of processing speed.
Flanker Task | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Flanker Task (FT) is a computerized assessment of selective attention and inhibitory control from the ExecQC Battery administered via Pavlovia. Participants identify the direction of a central arrow while ignoring flanking arrows that are either congruent (pointing same direction) or incongruent (pointing opposite direction) with the target. The primary outcome is the Flanker interference effect: the difference in reaction time between incongruent and congruent trials (lower = better inhibitory control). Additional outcomes include overall accuracy and congruency effect on accuracy. This task measures the ability to suppress irrelevant information and maintain attention on task-relevant stimuli.
Balloon Analogue Risk Task | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Balloon Analogue Risk Task (BART) is a computerized behavioral measure of risk-taking propensity and decision-making from the ExecQC Battery administered via Pavlovia. Participants inflate virtual balloons by pressing a key, earning points with each pump. Balloons have variable explosion points; if a balloon explodes, all points for that trial are lost. Participants can bank points at any time before explosion. The primary outcome is the adjusted average number of pumps on unexploded balloons, which reflects risk-taking behavior while controlling for random balloon explosion points. Higher scores indicate greater risk-taking. The task also yields measures of risk adjustment following losses and overall points earned.
Rey Auditory Verbal Learning Test | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Rey Auditory Verbal Learning Test (RAVLT) is a neuropsychological test measuring verbal memory and learning administered remotely via secure Zoom videoconferencing. The examiner reads a 15-word list (List A) aloud five times through the video platform, and the participant verbally recalls as many words as possible after each presentation. The Total Learning Score is the sum of correctly recalled words across all five trials, ranging from 0 to 75, with higher scores indicating better verbal learning and immediate memory. After a 20-minute delay filled with other cognitive tasks, participants are asked to verbally recall as many words as possible from the original list without re-presentation (Delayed Recall Score, range 0-15). Higher delayed recall scores indicate better long-term verbal memory and consolidation. This remote administration format has been validated for telehealth neuropsychological assessment and maintains the psychometric properties of in-person administration.
Symbol Digit Modalities Test | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Symbol Digit Modalities Test (SDMT) is a brief screening measure of processing speed, visual scanning, and sustained attention administered remotely via Zoom. Participants receive a paper copy of the test form with a key showing nine abstract symbols paired with digits 1-9 at the top, and rows of symbols below. On the examiner's verbal cue via video, participants write the corresponding digit below each symbol as quickly as possible for 90 seconds while the examiner monitors via video to ensure compliance. The score is the total number of correct symbol-digit pairings completed, with no penalty for errors. Scores typically range from 0 to approximately 110, with higher scores indicating faster processing speed. The written version is used for remote administration and has equivalent psychometric properties to oral administration.
Emotional Stroop Test | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Emotional Stroop Test measures selective attention and inhibitory control in the context of emotionally valenced stimuli, administered remotely via Zoom with stimuli presented through screen sharing. Participants view colored words displayed on the examiner's shared screen and verbally name the ink color while ignoring the word content. The test includes three conditions: neutral words (e.g., "table," "chair"), general emotional words (positive/negative: e.g., "happy," "angry"), and trauma-related words specific to PTSD (e.g., "danger," "threat"). Response latencies are recorded. The interference score is calculated by subtracting the mean reaction time for neutral words from the mean reaction time for trauma-related words. Higher interference scores (in milliseconds) indicate greater difficulty inhibiting attention to trauma-relevant content and poorer attentional control. Remote administration via screen sharing maintains the essential attentional demands of the task.
Verbal Fluency Test | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Verbal Fluency Test is a neuropsychological assessment measuring phonemic and semantic verbal fluency, executive functions, and language production administered remotely via Zoom. The test consists of two conditions: (1) Phonemic Fluency - participants generate as many words as possible beginning with the letter "P" in 90 seconds, excluding proper nouns and words from the same word family; and (2) Semantic Fluency - participants generate as many animal names as possible in 90 seconds, regardless of starting letter. The examiner monitors via video and records responses at 15-second intervals. Primary outcomes are the total number of correct responses in 60 seconds for each condition (typically ranging from 0 to 25+ words for phonemic and 0 to 30+ words for semantic).

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report questionnaire assessing PTSD symptom severity based on DSM-5 criteria. Participants rate how much they have been bothered by each PTSD symptom over the past month using a 5-point Likert scale (0 = Not at all, 1 = A little bit, 2 = Moderately, 3 = Quite a bit, 4 = Extremely). Total scores range from 0 to 80. Higher scores indicate greater PTSD symptom severity. A score of 33 or higher suggests probable PTSD diagnosis. The PCL-5 assesses four symptom clusters: intrusion symptoms, avoidance, negative alterations in cognitions and mood, and alterations in arousal and reactivity.
Patient Health Questionnaire-9 | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report questionnaire measuring depression severity based on DSM-5 criteria. Participants rate how often they have been bothered by depressive symptoms over the past two weeks using a 4-point scale (0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day). Total scores range from 0 to 27. Score interpretations: 0-4 (minimal depression), 5-9 (mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression), 20-27 (severe depression). Higher scores indicate greater depression severity.
Generalized Anxiety Disorder-7 | Baseline (Week 0), Post-intervention (Week 8), 3-month follow-up (Week 20)
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report questionnaire measuring generalized anxiety disorder symptom severity. Participants rate how often they have been bothered by anxiety symptoms over the past two weeks using a 4-point scale (0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day). Total scores range from 0 to 21. Score interpretations: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), 15-21 (severe anxiety). Higher scores indicate greater anxiety severity.
Strategy Use Questionnaire - Frequency of Strategy Application | 3-month follow-up only (Week 20)
  A brief questionnaire administered at 3-month follow-up assessing whether participants continued to apply cognitive strategies learned during the intervention. Participants indicate: (1) whether they have used any exercises or strategies since treatment completion (Yes/No), (2) if yes, the approximate number of times they have used them (0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, or 20+ times), and (3) an open-ended description of which specific strategies they have used. This measure captures maintenance of treatment effects and real-world application of learned compensatory strategies, which may mediate long-term outcomes.

OTHER OUTCOMES:
Weekly self-report of alcohol, drug, or non-prescribed medication use frequency | Weekly throughout 8-week intervention (Weeks 1-8)
  Participants complete a brief weekly questionnaire assessing substance use over the past week using a 4-point scale (0 = Never, 1 = A few days, 2 = More than half the days, 3 = Every day). This safety monitoring measure tracks potential increases in maladaptive coping behaviors during the intervention period. Significant increases in substance use may indicate treatment-related distress requiring clinical attention.
Weekly self-report of suicidal ideation frequency (PHQ-9 Item 9) | Weekly throughout 8-week intervention (Weeks 1-8)
  Participants complete PHQ-9 item 9 weekly, rating how often they have had thoughts that they would be better off dead or of hurting themselves over the past week using a 4-point scale (0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day). This safety monitoring measure tracks suicidal ideation throughout the intervention. Any positive response triggers the Columbia-Suicide Severity Rating Scale (C-SSRS) assessment to evaluate risk level and implement safety protocols as needed.
Weekly self-report of number of psychotherapy sessions attended | Weekly throughout 8-week intervention (Weeks 1-8)
  Participants report the number of psychotherapy sessions attended during the past week (0, 1, 2, 3, 4, or 5+ sessions). This measure tracks concurrent psychological treatment that may influence outcomes. Note: Cognitive remediation sessions are explicitly excluded from this count. This variable will be included as a covariate in outcome analyses to account for the potential additive or interactive effects of concurrent psychotherapy on cognitive and psychological outcomes.
Weekly self-report of any changes in psychiatric medications | Weekly throughout 8-week intervention (Weeks 1-8)
  Participants report any changes in psychiatric medications each week (Yes/No). If yes, they provide details about medication additions, discontinuations, or dose modifications, including medication names and dosages. This measure monitors potential medication changes that may influence treatment outcomes. Significant medication changes will be documented and considered in outcome analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Pavillon Adrien-Pinard (SU), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ainamani HE, Elbert T, Olema DK, Hecker T. PTSD symptom severity relates to cognitive and psycho-social dysfunctioning - a study with Congolese refugees in Uganda. Eur J Psychotraumatol. 2017 Feb 14;8(1):1283086. doi: 10.1080/20008198.2017.1283086. eCollection 2017. PMID 28326164
- [Background] Alioto AG, Kramer JH, Borish S, Neuhaus J, Saloner R, Wynn M, Foley JM. Long-term test-retest reliability of the California Verbal Learning Test - second edition. Clin Neuropsychol. 2017 Nov;31(8):1449-1458. doi: 10.1080/13854046.2017.1310300. Epub 2017 Apr 7. PMID 28387582
- [Background] Alon Y, Naim R, Pine DS, Bliese PD, Bar-Haim Y. Validity of Attention Bias Variability Indices for Posttraumatic Stress Disorder Research: Evidence From Patient Data. J Trauma Stress. 2019 Oct;32(5):791-798. doi: 10.1002/jts.22443. Epub 2019 Aug 28. PMID 31461560
- [Background] American Psychiatric Association. (2013). Diagnostic and Statistical Manual of Mental Disorders (5th ed.). Arlington, VA: American Psychiatric Publishing.
- [Background] Ashbaugh AR, Houle-Johnson S, Herbert C, El-Hage W, Brunet A. Psychometric Validation of the English and French Versions of the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). PLoS One. 2016 Oct 10;11(10):e0161645. doi: 10.1371/journal.pone.0161645. eCollection 2016. PMID 27723815
- [Background] Aupperle RL, Allard CB, Grimes EM, Simmons AN, Flagan T, Behrooznia M, Cissell SH, Twamley EW, Thorp SR, Norman SB, Paulus MP, Stein MB. Dorsolateral prefrontal cortex activation during emotional anticipation and neuropsychological performance in posttraumatic stress disorder. Arch Gen Psychiatry. 2012 Apr;69(4):360-71. doi: 10.1001/archgenpsychiatry.2011.1539. PMID 22474105
- [Background] Balzan RP, Mattiske JK, Delfabbro P, Liu D, Galletly C. Individualized Metacognitive Training (MCT+) Reduces Delusional Symptoms in Psychosis: A Randomized Clinical Trial. Schizophr Bull. 2019 Jan 1;45(1):27-36. doi: 10.1093/schbul/sby152. PMID 30376124
- [Background] Bandura, A. (1986). Social foundations of thought and action: A social cognitive theory. Englewood Cliffs, NJ: Prentice-Hall.
- [Background] Barlati S, Deste G, De Peri L, Ariu C, Vita A. Cognitive remediation in schizophrenia: current status and future perspectives. Schizophr Res Treatment. 2013;2013:156084. doi: 10.1155/2013/156084. Epub 2013 Dec 17. PMID 24455253
- [Background] Barrera, M. (1986). Distinctions between social support concepts, measures, and models. American Journal of Community Psychology, 14(4), 413-445. https://doi.org/10.1007/BF00922627
- [Background] Bates D, Mächler M, Bolker B, Walker S (2015). "Fitting Linear Mixed-Effects Models Using lme4." Journal of Statistical Software, 67(1), 1-48. doi:10.18637/jss.v067.i01.
- [Background] Baumann C, Erpelding ML, Regat S, Collin JF, Briancon S. The WHOQOL-BREF questionnaire: French adult population norms for the physical health, psychological health and social relationship dimensions. Rev Epidemiol Sante Publique. 2010 Feb;58(1):33-9. doi: 10.1016/j.respe.2009.10.009. Epub 2010 Jan 21. PMID 20096515
- [Background] Bayley MT, Janzen S, Harnett A, Teasell R, Patsakos E, Marshall S, Bragge P, Velikonja D, Kua A, Douglas J, Togher L, Ponsford J, McIntyre A. INCOG 2.0 Guidelines for Cognitive Rehabilitation Following Traumatic Brain Injury: Methods, Overview, and Principles. J Head Trauma Rehabil. 2023 Jan-Feb 01;38(1):7-23. doi: 10.1097/HTR.0000000000000838. PMID 36594856
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Belanger HG, Vanderploeg RD, Curtiss G, Armistead-Jehle P, Kennedy JE, Tate DF, Eapen BC, Bowles AO, Cooper DB. Self-efficacy predicts response to cognitive rehabilitation in military service members with post-concussive symptoms. Neuropsychol Rehabil. 2020 Jul;30(6):1190-1203. doi: 10.1080/09602011.2019.1575245. Epub 2019 Feb 15. PMID 30764711
- [Background] Best MW, Milanovic M, Tran T, Leung P, Jackowich R, Gauvin S, Leibovitz T, Bowie CR. Motivation and engagement during cognitive training for schizophrenia spectrum disorders. Schizophr Res Cogn. 2019 May 23;19:100151. doi: 10.1016/j.scog.2019.100151. eCollection 2020 Mar. PMID 31828022
- [Background] Bisson JI, Ehlers A, Matthews R, Pilling S, Richards D, Turner S. Psychological treatments for chronic post-traumatic stress disorder. Systematic review and meta-analysis. Br J Psychiatry. 2007 Feb;190:97-104. doi: 10.1192/bjp.bp.106.021402. PMID 17267924
- [Background] Bomyea J, Stein MB, Lang AJ. Interference control training for PTSD: A randomized controlled trial of a novel computer-based intervention. J Anxiety Disord. 2015 Aug;34:33-42. doi: 10.1016/j.janxdis.2015.05.010. Epub 2015 Jun 10. PMID 26114901
- [Background] Bongaerts H, Voorendonk EM, Van Minnen A, Rozendaal L, Telkamp BSD, de Jongh A. Fully remote intensive trauma-focused treatment for PTSD and Complex PTSD. Eur J Psychotraumatol. 2022 Sep 22;13(2):2103287. doi: 10.1080/20008066.2022.2103287. eCollection 2022. PMID 36186161
- [Background] Bouchard S, Bastien C, Morin CM. Self-efficacy and adherence to cognitive-behavioral treatment of insomnia. Behav Sleep Med. 2003;1(4):187-99. doi: 10.1207/S15402010BSM0104_2. PMID 15600214
- [Background] Boudrot, A., Sheehan, D., & Acquadro, C. (2013). Lost in Translation: Translatability of Psychiatric Terms - The Example of the Mini-International Neuropsychiatric Interview (M.I.N.I.). Value in Health, 16(7). https://doi.org/10.1016/j.jval.2013.08.1692
- [Background] Bowie CR. Cognitive remediation for severe mental illness: state of the field and future directions. World Psychiatry. 2019 Oct;18(3):274-275. doi: 10.1002/wps.20660. No abstract available. PMID 31496075
- [Background] Bowie CR, McGurk SR, Mausbach B, Patterson TL, Harvey PD. Combined cognitive remediation and functional skills training for schizophrenia: effects on cognition, functional competence, and real-world behavior. Am J Psychiatry. 2012 Jul;169(7):710-8. doi: 10.1176/appi.ajp.2012.11091337. PMID 22581070
- [Background] Boyd JE, O'Connor C, Protopopescu A, Jetly R, Rhind SG, Lanius RA, McKinnon MC. An Open-Label Feasibility Trial Examining the Effectiveness of a Cognitive Training Program, Goal Management Training, in Individuals With Posttraumatic Stress Disorder. Chronic Stress (Thousand Oaks). 2019 Apr 18;3:2470547019841599. doi: 10.1177/2470547019841599. eCollection 2019 Jan-Dec. PMID 32440592
- [Background] Boyer, P. (1996). L'Échelle d'Évaluation Globale de Fonctionnement (EGF). L'évaluation clinique standardisée en psychiatrie, tome 1. Éditions Pierre Fabre.
- [Background] Brandes D, Ben-Schachar G, Gilboa A, Bonne O, Freedman S, Shalev AY. PTSD symptoms and cognitive performance in recent trauma survivors. Psychiatry Res. 2002 Jul 31;110(3):231-8. doi: 10.1016/s0165-1781(02)00125-7. PMID 12127473
- [Background] Bremner JD, Randall P, Scott TM, Capelli S, Delaney R, McCarthy G, Charney DS. Deficits in short-term memory in adult survivors of childhood abuse. Psychiatry Res. 1995 Nov 29;59(1-2):97-107. doi: 10.1016/0165-1781(95)02800-5. PMID 8771224
- [Background] Bressan RA, Quarantini LC, Andreoli SB, Araujo C, Breen G, Guindalini C, Hoexter M, Jackowski AP, Jorge MR, Lacerda AL, Lara DR, Malta S, Moriyama TS, Quintana MI, Ribeiro WS, Ruiz J, Schoedl AF, Shih MC, Figueira I, Koenen KC, Mello MF, Mari JJ. The posttraumatic stress disorder project in Brazil: neuropsychological, structural and molecular neuroimaging studies in victims of urban violence. BMC Psychiatry. 2009 Jun 1;9:30. doi: 10.1186/1471-244X-9-30. PMID 19480721
- [Background] Campbell, T. A., PhD., Nelson, L. A., PhD., Lumpkin, R., B.A., Yoash-Gantz, R., Pickett, T. C., PsyD., & McCormick, C. L., M.A. (2009). Neuropsychological Measures of Processing Speed and Executive Functioning in Combat Veterans with PTSD, TBI, and Comorbid TBI/PTSD. Psychiatric Annals, 39(8), 796-803.
- [Background] Casada JH, Roache JD. Behavioral inhibition and activation in posttraumatic stress disorder. J Nerv Ment Dis. 2005 Feb;193(2):102-9. doi: 10.1097/01.nmd.0000152809.20938.37. PMID 15684912
- [Background] Choi J, Medalia A. Factors associated with a positive response to cognitive remediation in a community psychiatric sample. Psychiatr Serv. 2005 May;56(5):602-4. doi: 10.1176/appi.ps.56.5.602. PMID 15872171
- [Background] Cicerone KD, Goldin Y, Ganci K, Rosenbaum A, Wethe JV, Langenbahn DM, Malec JF, Bergquist TF, Kingsley K, Nagele D, Trexler L, Fraas M, Bogdanova Y, Harley JP. Evidence-Based Cognitive Rehabilitation: Systematic Review of the Literature From 2009 Through 2014. Arch Phys Med Rehabil. 2019 Aug;100(8):1515-1533. doi: 10.1016/j.apmr.2019.02.011. Epub 2019 Mar 26. PMID 30926291
- [Background] Clausen AN, Thelen J, Francisco AJ, Bruce J, Martin L, McDowd J, Aupperle RL. Computer-Based Executive Function Training for Combat Veterans With PTSD: A Pilot Clinical Trial Assessing Feasibility and Predictors of Dropout. Front Psychiatry. 2019 Mar 1;10:62. doi: 10.3389/fpsyt.2019.00062. eCollection 2019. PMID 30881315
- [Background] Cohen E, Zerach G, Solomon Z. The implication of combat-induced stress reaction, PTSD, and attachment in parenting among war veterans. J Fam Psychol. 2011 Oct;25(5):688-98. doi: 10.1037/a0024065. PMID 21639634
- [Background] Cohen, S., & Hoberman, H. M. (1983). Positive events and social supports as buffers of life change stress. Journal of Applied Social Psychology, 13(2), 99-125. https://doi.org/10.1111/j.1559-1816.1983.tb02325.x
- [Background] Conus P, Cotton S, Schimmelmann BG, Berk M, Daglas R, McGorry PD, Lambert M. Pretreatment and outcome correlates of past sexual and physical trauma in 118 bipolar I disorder patients with a first episode of psychotic mania. Bipolar Disord. 2010 May;12(3):244-52. doi: 10.1111/j.1399-5618.2010.00813.x. PMID 20565431
- [Background] Creamer M, Foran J, Bell R. The Beck Anxiety Inventory in a non-clinical sample. Behav Res Ther. 1995 May;33(4):477-85. doi: 10.1016/0005-7967(94)00082-u. PMID 7755538
- [Background] Delis, D. C., Kaplan, E., & Kramer, J. H. (2001). Delis Kaplan Executive Function System: Technical Manual. San Antonio: The Psychological Corporation.
- [Background] Delis, D. C., Kramer, J. H., Kaplan, E., & Ober, B. A. (1987-2000). California Verbal Learning Test--Second Edition (CVLT -II) [Database record]. APA PsycTests. https://doi.org/10.1037/t15072-000
- [Background] Denis A, Callahan S, Bouvard M. Evaluation of the French version of the multidimensional scale of perceived social support during the postpartum period. Matern Child Health J. 2015 Jun;19(6):1245-51. doi: 10.1007/s10995-014-1630-9. PMID 25366102
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Dumont, M., Schwarzer, R., & Jerusalem, M. (2000). French Adaptation of the General Self-Efficacy Scale. Retrieved August 28, 2022, from http://userpage.fu-berlin.de/~health/french.htm
- [Background] Dutra SJ, Marx BP, McGlinchey R, DeGutis J, Esterman M. Reward Ameliorates Posttraumatic Stress Disorder-Related Impairment in Sustained Attention. Chronic Stress (Thousand Oaks). 2018 Jan-Dec;2:2470547018812400. doi: 10.1177/2470547018812400. Epub 2018 Nov 26. PMID 30706031
- [Background] Eichner C, Berna F. Acceptance and Efficacy of Metacognitive Training (MCT) on Positive Symptoms and Delusions in Patients With Schizophrenia: A Meta-analysis Taking Into Account Important Moderators. Schizophr Bull. 2016 Jul;42(4):952-62. doi: 10.1093/schbul/sbv225. Epub 2016 Jan 8. PMID 26748396
- [Background] Esterman M, Reagan A, Liu G, Turner C, DeGutis J. Reward reveals dissociable aspects of sustained attention. J Exp Psychol Gen. 2014 Dec;143(6):2287-95. doi: 10.1037/xge0000019. Epub 2014 Oct 13. PMID 25313950
- [Background] Esterman M, Rothlein D. Models of sustained attention. Curr Opin Psychol. 2019 Oct;29:174-180. doi: 10.1016/j.copsyc.2019.03.005. Epub 2019 Mar 13. PMID 30986621
- [Background] Falconer E, Bryant R, Felmingham KL, Kemp AH, Gordon E, Peduto A, Olivieri G, Williams LM. The neural networks of inhibitory control in posttraumatic stress disorder. J Psychiatry Neurosci. 2008 Sep;33(5):413-22. PMID 18787658
- [Background] Fioravanti M, Carlone O, Vitale B, Cinti ME, Clare L. A meta-analysis of cognitive deficits in adults with a diagnosis of schizophrenia. Neuropsychol Rev. 2005 Jun;15(2):73-95. doi: 10.1007/s11065-005-6254-9. PMID 16211467
- [Background] Fletcher S, Elklit A, Shevlin M, Armour C. Predictors of PTSD Treatment Response Trajectories in a Sample of Childhood Sexual Abuse Survivors: The Roles of Social Support, Coping, and PTSD Symptom Clusters. J Interpers Violence. 2021 Feb;36(3-4):1283-1307. doi: 10.1177/0886260517741212. Epub 2017 Nov 15. PMID 29294985
- [Background] Foa E. B., Keane T. M., Friedman M. J., Cohen J. A. (2009). Effective Treatments for PTSD: Practice Guidelines from the International Society for Traumatic Stress Studies. 2nd Edn. New York, NY: The Guilford Press.
- [Background] Fonzo GA, Fine NB, Wright RN, Achituv M, Zaiko YV, Merin O, Shalev AY, Etkin A. Internet-delivered computerized cognitive & affective remediation training for the treatment of acute and chronic posttraumatic stress disorder: Two randomized clinical trials. J Psychiatr Res. 2019 Aug;115:82-89. doi: 10.1016/j.jpsychires.2019.05.007. Epub 2019 May 8. PMID 31125916
- [Background] Fortenbaugh FC, Corbo V, Poole V, McGlinchey R, Milberg W, Salat D, DeGutis J, Esterman M. Interpersonal early-life trauma alters amygdala connectivity and sustained attention performance. Brain Behav. 2017 Apr 10;7(5):e00684. doi: 10.1002/brb3.684. eCollection 2017 May. PMID 28523226
- [Background] Gallagher MW, Payne LA, White KS, Shear KM, Woods SW, Gorman JM, Barlow DH. Mechanisms of change in cognitive behavioral therapy for panic disorder: the unique effects of self-efficacy and anxiety sensitivity. Behav Res Ther. 2013 Nov;51(11):767-77. doi: 10.1016/j.brat.2013.09.001. Epub 2013 Sep 12. PMID 24095901
- [Background] Geuze E, Vermetten E, de Kloet CS, Hijman R, Westenberg HG. Neuropsychological performance is related to current social and occupational functioning in veterans with posttraumatic stress disorder. Depress Anxiety. 2009;26(1):7-15. doi: 10.1002/da.20476. PMID 18800372
- [Background] Gold JM, Goldberg RW, McNary SW, Dixon LB, Lehman AF. Cognitive correlates of job tenure among patients with severe mental illness. Am J Psychiatry. 2002 Aug;159(8):1395-402. doi: 10.1176/appi.ajp.159.8.1395. PMID 12153834
- [Background] Green MF, Kern RS, Braff DL, Mintz J. Neurocognitive deficits and functional outcome in schizophrenia: are we measuring the "right stuff"? Schizophr Bull. 2000;26(1):119-36. doi: 10.1093/oxfordjournals.schbul.a033430. PMID 10755673
- [Background] Grynszpan O, Perbal S, Pelissolo A, Fossati P, Jouvent R, Dubal S, Perez-Diaz F. Efficacy and specificity of computer-assisted cognitive remediation in schizophrenia: a meta-analytical study. Psychol Med. 2011 Jan;41(1):163-73. doi: 10.1017/S0033291710000607. Epub 2010 Apr 12. PMID 20380784
- [Background] Harris AW, Kosic T, Xu J, Walker C, Gye W, Redoblado Hodge A. Web-Based Cognitive Remediation Improves Supported Employment Outcomes in Severe Mental Illness: Randomized Controlled Trial. JMIR Ment Health. 2017 Sep 20;4(3):e30. doi: 10.2196/mental.6982. PMID 28931500
- [Background] Hayes, A. F. (2022). Introduction to mediation, moderation, and conditional process analysis: A regression-based approach. Third edition. Guilford publications.
- [Background] Heaton, R. K. (1993). Wisconsin Card Sorting Test Manual: Revised and expanded. Psychological Assessment Resources.
- [Background] Hilsenroth MJ, Ackerman SJ, Blagys MD, Baumann BD, Baity MR, Smith SR, Price JL, Smith CL, Heindselman TL, Mount MK, Holdwick DJ Jr. Reliability and validity of DSM-IV axis V. Am J Psychiatry. 2000 Nov;157(11):1858-63. doi: 10.1176/appi.ajp.157.11.1858. PMID 11058486
- [Background] Horner MD, Hamner MB. Neurocognitive functioning in posttraumatic stress disorder. Neuropsychol Rev. 2002 Mar;12(1):15-30. doi: 10.1023/a:1015439106231. PMID 12090717
- [Background] Jagtap S, Romanowska S, Leibovitz T, Onno KA, Burhan AM, Best MW. Can cognitive remediation therapy be delivered remotely? A review examining feasibility and acceptability of remote interventions. Schizophr Res Cogn. 2022 Jan 25;28:100238. doi: 10.1016/j.scog.2022.100238. eCollection 2022 Jun. PMID 35242607
- [Background] Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials - a practical guide with flowcharts. BMC Med Res Methodol. 2017 Dec 6;17(1):162. doi: 10.1186/s12874-017-0442-1. PMID 29207961
- [Background] Jenkins MA, Langlais PJ, Delis DA, Cohen RA. Attentional dysfunction associated with posttraumatic stress disorder among rape survivors. Clin Neuropsychol. 2000 Feb;14(1):7-12. doi: 10.1076/1385-4046(200002)14:1;1-8;FT007. PMID 10855055
- [Background] Jenkins MA, Langlais PJ, Delis D, Cohen R. Learning and memory in rape victims with posttraumatic stress disorder. Am J Psychiatry. 1998 Feb;155(2):278-9. doi: 10.1176/ajp.155.2.278. PMID 9464211
- [Background] Johnsen GE, Asbjornsen AE. Consistent impaired verbal memory in PTSD: a meta-analysis. J Affect Disord. 2008 Nov;111(1):74-82. doi: 10.1016/j.jad.2008.02.007. Epub 2008 Apr 2. PMID 18377999
- [Background] Jun J, Lee VG. Perceptual and response factors in the gradual onset continuous performance tasks. Atten Percept Psychophys. 2021 Oct;83(7):3008-3023. doi: 10.3758/s13414-021-02353-7. Epub 2021 Aug 5. PMID 34355343
- [Background] Kalechstein AD, Newton TF, van Gorp WG. Neurocognitive functioning is associated with employment status: a quantitative review. J Clin Exp Neuropsychol. 2003 Dec;25(8):1186-91. doi: 10.1076/jcen.25.8.1186.16723. PMID 14566590
- [Background] Kanagaratnam P, Asbjornsen AE. Executive deficits in chronic PTSD related to political violence. J Anxiety Disord. 2007;21(4):510-25. doi: 10.1016/j.janxdis.2006.06.008. Epub 2006 Aug 30. PMID 16938424
- [Background] Kavanagh DJ, Wilson PH. Prediction of outcome with group cognitive therapy for depression. Behav Res Ther. 1989;27(4):333-43. doi: 10.1016/0005-7967(89)90003-x. PMID 2775143
- [Background] Kar N. Cognitive behavioral therapy for the treatment of post-traumatic stress disorder: a review. Neuropsychiatr Dis Treat. 2011;7:167-81. doi: 10.2147/NDT.S10389. Epub 2011 Apr 4. PMID 21552319
- [Background] Keane TM, Kaloupek DG. Imaginal flooding in the treatment of a posttraumatic stress disorder. J Consult Clin Psychol. 1982 Feb;50(1):138-40. doi: 10.1037//0022-006x.50.1.138. No abstract available. PMID 7056906
- [Background] Keshavan MS, Vinogradov S, Rumsey J, Sherrill J, Wagner A. Cognitive training in mental disorders: update and future directions. Am J Psychiatry. 2014 May;171(5):510-22. doi: 10.1176/appi.ajp.2013.13081075. PMID 24700194
- [Background] Keshen A, Helson T, Town J, Warren K. Self-efficacy as a predictor of treatment outcome in an outpatient eating disorder program. Eat Disord. 2017 Oct-Dec;25(5):406-419. doi: 10.1080/10640266.2017.1324073. Epub 2017 May 12. PMID 28498014
- [Background] Kessler RC. Posttraumatic stress disorder: the burden to the individual and to society. J Clin Psychiatry. 2000;61 Suppl 5:4-12; discussion 13-4. PMID 10761674
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Kim EJ, Bahk YC, Oh H, Lee WH, Lee JS, Choi KH. Current Status of Cognitive Remediation for Psychiatric Disorders: A Review. Front Psychiatry. 2018 Oct 1;9:461. doi: 10.3389/fpsyt.2018.00461. eCollection 2018. PMID 30337888
- [Background] Koso M, Hansen S. Executive function and memory in posttraumatic stress disorder: a study of Bosnian war veterans. Eur Psychiatry. 2006 Apr;21(3):167-73. doi: 10.1016/j.eurpsy.2005.06.004. Epub 2005 Aug 31. PMID 16139487
- [Background] Kurtz, M. M. (2016). Cognitive remediation for psychological disorders: An overview. In A. Medalia & C. R. Bowie (Eds.), Cognitive remediation to improve functional outcomes (pp. 1-23). Oxford University Press. https://doi.org/10.1093/med:psych/9780199395224.003.0001
- [Background] Kurtz MM, Moberg PJ, Gur RC, Gur RE. Approaches to cognitive remediation of neuropsychological deficits in schizophrenia: a review and meta-analysis. Neuropsychol Rev. 2001 Dec;11(4):197-210. doi: 10.1023/a:1012953108158. PMID 11883669
- [Background] Lagarde G, Doyon J, Brunet A. Memory and executive dysfunctions associated with acute posttraumatic stress disorder. Psychiatry Res. 2010 May 15;177(1-2):144-9. doi: 10.1016/j.psychres.2009.02.002. Epub 2010 Apr 9. PMID 20381880
- [Background] Langner R, Eickhoff SB. Sustaining attention to simple tasks: a meta-analytic review of the neural mechanisms of vigilant attention. Psychol Bull. 2013 Jul;139(4):870-900. doi: 10.1037/a0030694. Epub 2012 Nov 19. PMID 23163491
- [Background] Lavigne KM, Sauve G, Raucher-Chene D, Guimond S, Lecomte T, Bowie CR, Menon M, Lal S, Woodward TS, Bodnar MD, Lepage M. Remote cognitive assessment in severe mental illness: a scoping review. Schizophrenia (Heidelb). 2022 Mar 5;8(1):14. doi: 10.1038/s41537-022-00219-x. PMID 35249112
- [Background] Lecrubier, Y., Sheehan, D. V., Weiller, E., Amorim, P., Bonora, I., Sheehan, K. H., Janavs, J., & Dunbar, G. C. (1997). The Mini International Neuropsychiatric Interview (MINI). A short diagnostic structured interview: reliability and validity according to the CIDI. European Psychiatry, 12(5), 224-231.
- [Background] Leskin LP, White PM. Attentional networks reveal executive function deficits in posttraumatic stress disorder. Neuropsychology. 2007 May;21(3):275-84. doi: 10.1037/0894-4105.21.3.275. PMID 17484590
- [Background] Lindauer RJ, Olff M, van Meijel EP, Carlier IV, Gersons BP. Cortisol, learning, memory, and attention in relation to smaller hippocampal volume in police officers with posttraumatic stress disorder. Biol Psychiatry. 2006 Jan 15;59(2):171-7. doi: 10.1016/j.biopsych.2005.06.033. Epub 2005 Sep 9. PMID 16154543
- [Background] Lindenmayer JP, Ozog VA, Khan A, Ljuri I, Fregenti S, McGurk SR. Predictors of response to cognitive remediation in service recipients with severe mental illness. Psychiatr Rehabil J. 2017 Mar;40(1):61-69. doi: 10.1037/prj0000252. PMID 28368180
- [Background] Lowe C, Rabbitt P. Test/re-test reliability of the CANTAB and ISPOCD neuropsychological batteries: theoretical and practical issues. Cambridge Neuropsychological Test Automated Battery. International Study of Post-Operative Cognitive Dysfunction. Neuropsychologia. 1998 Sep;36(9):915-23. doi: 10.1016/s0028-3932(98)00036-0. PMID 9740364
- [Background] McGurk, S. R., & Mueser, K. T. (2008). Response to cognitive rehabilitation in older versus younger persons with severe mental illness. American Journal of Psychiatric Rehabilitation, 11(1), 90-105.
- [Background] Medalia, A. and Freilich, B. (2008) The Neuropsychological Educational Approach to Cognitive Remediation (NEAR) Model: Practice Principles and Outcome Studies. American Journal of Psychiatric Rehabilitation, 11, 23-143. https://doi.org/10.1080/15487760801963660
- [Background] Medalia A, Richardson R. What predicts a good response to cognitive remediation interventions? Schizophr Bull. 2005 Oct;31(4):942-53. doi: 10.1093/schbul/sbi045. Epub 2005 Aug 24. PMID 16120830
- [Background] Medalia A, Saperstein AM. Does cognitive remediation for schizophrenia improve functional outcomes? Curr Opin Psychiatry. 2013 Mar;26(2):151-7. doi: 10.1097/YCO.0b013e32835dcbd4. PMID 23318663
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] Mendelson D, Thibaudeau E, Sauve G, Lavigne KM, Bowie CR, Menon M, Woodward TS, Lepage M, Raucher-Chene D. Remote group therapies for cognitive health in schizophrenia-spectrum disorders: Feasible, acceptable, engaging. Schizophr Res Cogn. 2021 Dec 6;28:100230. doi: 10.1016/j.scog.2021.100230. eCollection 2022 Jun. PMID 35242604
- [Background] Miskowiak KW, Moller AB, Ott CV. Neuronal and cognitive predictors of improved executive function following action-based cognitive remediation in patients with bipolar disorder. Eur Neuropsychopharmacol. 2021 Jun;47:1-10. doi: 10.1016/j.euroneuro.2021.02.013. Epub 2021 Mar 13. PMID 33725651
- [Background] Mordal J, Gundersen O, Bramness JG. Norwegian version of the Mini-International Neuropsychiatric Interview: feasibility, acceptability and test-retest reliability in an acute psychiatric ward. Eur Psychiatry. 2010 Apr;25(3):172-7. doi: 10.1016/j.eurpsy.2009.02.004. Epub 2009 Jun 23. PMID 19553089
- [Background] Morosini PL, Magliano L, Brambilla L, Ugolini S, Pioli R. Development, reliability and acceptability of a new version of the DSM-IV Social and Occupational Functioning Assessment Scale (SOFAS) to assess routine social functioning. Acta Psychiatr Scand. 2000 Apr;101(4):323-9. PMID 10782554
- [Background] Motter JN, Pimontel MA, Rindskopf D, Devanand DP, Doraiswamy PM, Sneed JR. Computerized cognitive training and functional recovery in major depressive disorder: A meta-analysis. J Affect Disord. 2016 Jan 1;189:184-91. doi: 10.1016/j.jad.2015.09.022. Epub 2015 Sep 26. PMID 26437233
- [Background] Nijdam MJ, Gersons BP, Reitsma JB, de Jongh A, Olff M. Brief eclectic psychotherapy v. eye movement desensitisation and reprocessing therapy for post-traumatic stress disorder: randomised controlled trial. Br J Psychiatry. 2012 Mar;200(3):224-31. doi: 10.1192/bjp.bp.111.099234. Epub 2012 Feb 9. PMID 22322458
- [Background] Nolin, P. (1999). Analyses psychométriques de l'adaptation française du California Verbal Learning Test (CVLT). Revue québécoise de psychologie, 20(1), 39-55.
- [Background] Norman SB, Stein MB, Davidson JR. Profiling posttraumatic functional impairment. J Nerv Ment Dis. 2007 Jan;195(1):48-53. doi: 10.1097/01.nmd.0000252135.25114.02. PMID 17220739
- [Background] Olff M, Polak AR, Witteveen AB, Denys D. Executive function in posttraumatic stress disorder (PTSD) and the influence of comorbid depression. Neurobiol Learn Mem. 2014 Jul;112:114-21. doi: 10.1016/j.nlm.2014.01.003. Epub 2014 Jan 16. PMID 24440596
- [Background] Oquendo, M.A. & Halberstam, B. & Mann, J. (2003). Risk factors for suicidal behavior. The utility and limitations of research instruments. Standardized Evaluation in Clinical Practice. Review of Psychiatry. 8. 103-130.
- [Background] Otsubo T, Tanaka K, Koda R, Shinoda J, Sano N, Tanaka S, Aoyama H, Mimura M, Kamijima K. Reliability and validity of Japanese version of the Mini-International Neuropsychiatric Interview. Psychiatry Clin Neurosci. 2005 Oct;59(5):517-26. doi: 10.1111/j.1440-1819.2005.01408.x. PMID 16194252
- [Background] Ott CV, Vinberg M, Kessing LV, Bowie CR, Forman JL, Miskowiak KW. Effect of Action-Based Cognitive Remediation on cognitive impairment in patients with remitted bipolar disorder: A randomized controlled trial. Bipolar Disord. 2021 Aug;23(5):487-499. doi: 10.1111/bdi.13021. Epub 2020 Oct 29. PMID 33053258
- [Background] Ozer EJ, Best SR, Lipsey TL, Weiss DS. Predictors of posttraumatic stress disorder and symptoms in adults: a meta-analysis. Psychol Bull. 2003 Jan;129(1):52-73. doi: 10.1037/0033-2909.129.1.52. PMID 12555794
- [Background] Palumbo D, Mucci A, Giordano GM, Piegari G, Aiello C, Pietrafesa D, Annarumma N, Chieffi M, Cella M, Galderisi S. The Efficacy, Feasibility And Acceptability Of A Remotely Accessible Use Of CIRCuiTS, A Computerized Cognitive Remediation Therapy Program For Schizophrenia: A Pilot Study. Neuropsychiatr Dis Treat. 2019 Nov 8;15:3103-3113. doi: 10.2147/NDT.S221690. eCollection 2019. PMID 31814722
- [Background] Pfizer (n.d.). Patient Health Questionnaire Screeners. https://www.phqscreeners.com/selectscreener
- [Background] Pinninti NR, Madison H, Musser E, Rissmiller D. MINI International Neuropsychiatric Schedule: clinical utility and patient acceptance. Eur Psychiatry. 2003 Nov;18(7):361-4. doi: 10.1016/j.eurpsy.2003.03.004. PMID 14643565
- [Background] Polak AR, Witteveen AB, Reitsma JB, Olff M. The role of executive function in posttraumatic stress disorder: a systematic review. J Affect Disord. 2012 Dec 1;141(1):11-21. doi: 10.1016/j.jad.2012.01.001. Epub 2012 Feb 5. PMID 22310036
- [Background] Ponniah K, Hollon SD. Empirically supported psychological treatments for adult acute stress disorder and posttraumatic stress disorder: a review. Depress Anxiety. 2009;26(12):1086-109. doi: 10.1002/da.20635. PMID 19957280
- [Background] Posner MI, Petersen SE. The attention system of the human brain. Annu Rev Neurosci. 1990;13:25-42. doi: 10.1146/annurev.ne.13.030190.000325. No abstract available. PMID 2183676
- [Background] Prikken M, Konings MJ, Lei WU, Begemann MJH, Sommer IEC. The efficacy of computerized cognitive drill and practice training for patients with a schizophrenia-spectrum disorder: A meta-analysis. Schizophr Res. 2019 Feb;204:368-374. doi: 10.1016/j.schres.2018.07.034. Epub 2018 Aug 7. PMID 30097278
- [Background] Rapaport MH, Clary C, Fayyad R, Endicott J. Quality-of-life impairment in depressive and anxiety disorders. Am J Psychiatry. 2005 Jun;162(6):1171-8. doi: 10.1176/appi.ajp.162.6.1171. PMID 15930066
- [Background] Robbins TW, James M, Owen AM, Sahakian BJ, Lawrence AD, McInnes L, Rabbitt PM. A study of performance on tests from the CANTAB battery sensitive to frontal lobe dysfunction in a large sample of normal volunteers: implications for theories of executive functioning and cognitive aging. Cambridge Neuropsychological Test Automated Battery. J Int Neuropsychol Soc. 1998 Sep;4(5):474-90. doi: 10.1017/s1355617798455073. PMID 9745237
- [Background] Rodriguez P, Holowka DW, Marx BP. Assessment of posttraumatic stress disorder-related functional impairment: a review. J Rehabil Res Dev. 2012;49(5):649-65. doi: 10.1682/jrrd.2011.09.0162. PMID 23015577
- [Background] Rossi A, Alberio R, Porta A, Sandri M, Tansella M, Amaddeo F. The reliability of the Mini-International Neuropsychiatric Interview--Italian version. J Clin Psychopharmacol. 2004 Oct;24(5):561-3. doi: 10.1097/01.jcp.0000139758.03834.ad. No abstract available. PMID 15349020
- [Background] Sachinvala N, von Scotti H, McGuire M, Fairbanks L, Bakst K, McGuire M, Fairbanks L, Bakst K, McGuire M, Brown N. Memory, attention, function, and mood among patients with chronic posttraumatic stress disorder. J Nerv Ment Dis. 2000 Dec;188(12):818-23. doi: 10.1097/00005053-200012000-00005. PMID 11191582
- [Background] Samuelson KW, Engle K, Bartel A, Jordan JT, Powers T, Abadjian L, Benight CC. The power of appraisals in predicting PTSD symptom improvement following cognitive rehabilitation: A randomized clinical trial. J Affect Disord. 2021 Mar 1;282:561-573. doi: 10.1016/j.jad.2020.12.067. Epub 2020 Dec 24. PMID 33440301
- [Background] Saunders N, Downham R, Turman B, Kropotov J, Clark R, Yumash R, Szatmary A. Working memory training with tDCS improves behavioral and neurophysiological symptoms in pilot group with post-traumatic stress disorder (PTSD) and with poor working memory. Neurocase. 2015;21(3):271-8. doi: 10.1080/13554794.2014.890727. Epub 2014 Feb 28. PMID 24579831
- [Background] Sautter FJ, Glynn SM, Thompson KE, Franklin L, Han X. A couple-based approach to the reduction of PTSD avoidance symptoms: preliminary findings. J Marital Fam Ther. 2009 Jul;35(3):343-9. doi: 10.1111/j.1752-0606.2009.00125.x. PMID 19522786
- [Background] Scholz, U., Doña, B. G., Sud, S., & Schwarzer, R. (2002). Is general self-efficacy a universal construct? Psychometric findings from 25 countries. European Journal of Psychological Assessment, 18(3), 242-251. https://doi.org/10.1027/1015-5759.18.3.242
- [Background] Schonning A, Nordgreen T. Predicting Treatment Outcomes in Guided Internet-Delivered Therapy for Anxiety Disorders-The Role of Treatment Self-Efficacy. Front Psychol. 2021 Oct 21;12:712421. doi: 10.3389/fpsyg.2021.712421. eCollection 2021. PMID 34744872
- [Background] Schulz-Heik RJ, Fahimi A, Durazzo TC, Friedman M, Bayley PJ. Evaluation of adding the CANTAB computerized neuropsychological assessment battery to a traditional battery in a tertiary care center for veterans. Appl Neuropsychol Adult. 2020 May-Jun;27(3):256-266. doi: 10.1080/23279095.2018.1534735. Epub 2019 Jan 11. PMID 30633552
- [Background] Schwarzer, R., & Jerusalem, M. (1995). General self-efficacy scale. PsycTESTS Dataset. https://doi.org/10.1037/t00393-000
- [Background] Schwarzer, R., & Knoll, N. (2007). Functional roles of social support within the stress and coping process: A theoretical and empirical overview. International Journal of Psychology, 42, 243-252. doi:10.1080/00207590701396641
- [Background] Scott JC, Matt GE, Wrocklage KM, Crnich C, Jordan J, Southwick SM, Krystal JH, Schweinsburg BC. A quantitative meta-analysis of neurocognitive functioning in posttraumatic stress disorder. Psychol Bull. 2015 Jan;141(1):105-140. doi: 10.1037/a0038039. Epub 2014 Nov 3. PMID 25365762
- [Background] Seccomandi B, Agbedjro D, Keefe RSE, Galderisi S, Fiszdon J, Mucci A, Wykes T, Cella M. Evaluating how treatment adherence influences cognitive remediation outcomes. Behav Res Ther. 2022 Nov;158:104186. doi: 10.1016/j.brat.2022.104186. Epub 2022 Aug 27. PMID 36096075
- [Background] Seccomandi B, Tsapekos D, Newbery K, Wykes T, Cella M. A systematic review of moderators of cognitive remediation response for people with schizophrenia. Schizophr Res Cogn. 2019 Sep 5;19:100160. doi: 10.1016/j.scog.2019.100160. eCollection 2020 Mar. PMID 31828023
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Sheehan, D.V., Lecrubier, Y., Sheehan, K. H., Janavs, J., Weiller, E., Keskiner, A., Schinka, J., Knapp, E., Sheehan, M. F., & Dunbar, G. C. (1997). The validity of the Mini International Neuropsychiatric Interview (MINI) according to the SCID-P and its reliability. European Psychiatry, 12(5), 232-241. https://doi.org/10.1016/S0924-9338(97)83297-X
- [Background] Shinn, M., Lehmann, S., & Wong, N. W. (1984). Social interaction and social support. Journal of Social Issues, 40(4), 55-76. https://doi.org/10.1111/j.1540-4560.1984.tb01107.x
- [Background] Shucard JL, McCabe DC, Szymanski H. An event-related potential study of attention deficits in posttraumatic stress disorder during auditory and visual Go/NoGo continuous performance tasks. Biol Psychol. 2008 Oct;79(2):223-33. doi: 10.1016/j.biopsycho.2008.05.005. Epub 2008 Jun 10. PMID 18590795
- [Background] Silverberg ND, Wojtowicz M, Bui E, Wershba R, Zafonte R, Laifer LM, Simon NM, Iverson GL. Contribution of Perceived Cognitive Functioning to Quality of Life in Service Members and Veterans With Posttraumatic Stress Disorder. J Trauma Stress. 2017 Jun;30(3):318-322. doi: 10.1002/jts.22184. Epub 2017 May 19. PMID 28544024
- [Background] Simon, H. A. (1975). The functional equivalence of problem solving skills. Cognitive Psychology, 7(2), 268-288. https://doi.org/10.1016/0010-0285(75)90012-2
- [Background] Snijders, T. A. (2005). Power and sample size in multilevel linear models. Encyclopedia of Statistics in Behavioral Science. https://doi.org/10.1002/0470013192.bsa492
- [Background] Solomon Z, Dekel R, Zerach G. The relationships between posttraumatic stress symptom clusters and marital intimacy among war veterans. J Fam Psychol. 2008 Oct;22(5):659-66. doi: 10.1037/a0013596. PMID 18855502
- [Background] Sonuga-Barke EJ, Brandeis D, Cortese S, Daley D, Ferrin M, Holtmann M, Stevenson J, Danckaerts M, van der Oord S, Dopfner M, Dittmann RW, Simonoff E, Zuddas A, Banaschewski T, Buitelaar J, Coghill D, Hollis C, Konofal E, Lecendreux M, Wong IC, Sergeant J; European ADHD Guidelines Group. Nonpharmacological interventions for ADHD: systematic review and meta-analyses of randomized controlled trials of dietary and psychological treatments. Am J Psychiatry. 2013 Mar;170(3):275-89. doi: 10.1176/appi.ajp.2012.12070991. PMID 23360949
- [Background] Statistiques Canada. (2021). Survey on Mental Health and Stressful Events, August to December 2021. (no. 11-001-X)
- [Background] Stein MB, Kennedy CM, Twamley EW. Neuropsychological function in female victims of intimate partner violence with and without posttraumatic stress disorder. Biol Psychiatry. 2002 Dec 1;52(11):1079-88. doi: 10.1016/s0006-3223(02)01414-2. PMID 12460691
- [Background] Susanty E, Sijbrandij M, van Dijk W, Srisayekti W, de Vries R, Huizink AC. The effects of psychological interventions on neurocognitive functioning in posttraumatic stress disorder: a systematic review. Eur J Psychotraumatol. 2022 May 26;13(1):2071527. doi: 10.1080/20008198.2022.2071527. eCollection 2022. PMID 35957628
- [Background] Swick D, Honzel N, Larsen J, Ashley V. Increased response variability as a marker of executive dysfunction in veterans with post-traumatic stress disorder. Neuropsychologia. 2013 Dec;51(14):3033-40. doi: 10.1016/j.neuropsychologia.2013.10.008. Epub 2013 Oct 21. PMID 24157540
- [Background] Swick D, Honzel N, Turken U. Intact error monitoring in combat Veterans with post-traumatic stress disorder. Psychiatry Res. 2015 Nov 30;234(2):227-38. doi: 10.1016/j.pscychresns.2015.09.016. Epub 2015 Sep 21. PMID 26481979
- [Background] Tedim Cruz V, Pais J, Alves I, Ruano L, Mateus C, Barreto R, Bento V, Colunas M, Rocha N, Coutinho P. Web-based cognitive training: patient adherence and intensity of treatment in an outpatient memory clinic. J Med Internet Res. 2014 May 7;16(5):e122. doi: 10.2196/jmir.3377. PMID 24808451
- [Background] Theofilou, P. (2013). RETRACTED: Quality of Life: Definition and Measurement. Europe's Journal of Psychology, 9(1), 150-162. https://doi.org/10.5964/ejop.v9i1.337 More Citation Formats
- [Background] Therond A, Pezzoli P, Abbas M, Howard A, Bowie CR, Guimond S. The Efficacy of Cognitive Remediation in Depression: A Systematic Literature Review and Meta-Analysis. J Affect Disord. 2021 Apr 1;284:238-246. doi: 10.1016/j.jad.2021.02.009. Epub 2021 Feb 9. PMID 33631438
- [Background] Thoits PA. Stress, coping, and social support processes: where are we? What next? J Health Soc Behav. 1995;Spec No:53-79. PMID 7560850
- [Background] Thrasher S, Power M, Morant N, Marks I, Dalgleish T. Social support moderates outcome in a randomized controlled trial of exposure therapy and (or) cognitive restructuring for chronic posttraumatic stress disorder. Can J Psychiatry. 2010 Mar;55(3):187-90. doi: 10.1177/070674371005500311. PMID 20370970
- [Background] Tsapekos D, Strawbridge R, Wykes T, Young AH, Cella M. Cognitive remediation for people with bipolar disorder: The contribution of session attendance and therapy components to cognitive and functional outcomes. J Psychiatr Res. 2022 Aug;152:144-151. doi: 10.1016/j.jpsychires.2022.06.021. Epub 2022 Jun 11. PMID 35724496
- [Background] Twamley EW, Allard CB, Thorp SR, Norman SB, Hami Cissell S, Hughes Berardi K, Grimes EM, Stein MB. Cognitive impairment and functioning in PTSD related to intimate partner violence. J Int Neuropsychol Soc. 2009 Nov;15(6):879-87. doi: 10.1017/S135561770999049X. Epub 2009 Aug 25. PMID 19703324
- [Background] Twamley EW, Jeste DV, Bellack AS. A review of cognitive training in schizophrenia. Schizophr Bull. 2003;29(2):359-82. doi: 10.1093/oxfordjournals.schbul.a007011. PMID 14552510
- [Background] Uddo, M., Vasterling, J. J., Brailey, K., & Sutker, P. B. (1993). Memory and attention in combat-related post-traumatic stress disorder (PTSD). Journal of Psychopathology and Behavioral Assessment, 15(1), 43-52. https://doi.org/10.1007/BF00964322
- [Background] Vasterling, J. J., & Brailey, K. (2005). Neuropsychological Findings in Adults with PTSD. In J. J.
- [Background] Vasterling & C. R. Brewin (Eds.), Neuropsychology of PTSD: Biological, cognitive, and clinical perspectives (pp. 178-207). The Guilford Press.
- [Background] Vasterling JJ, Brailey K, Constans JI, Sutker PB. Attention and memory dysfunction in posttraumatic stress disorder. Neuropsychology. 1998 Jan;12(1):125-33. doi: 10.1037//0894-4105.12.1.125. PMID 9460740
- [Background] Vasterling JJ, Duke LM, Brailey K, Constans JI, Allain AN Jr, Sutker PB. Attention, learning, and memory performances and intellectual resources in Vietnam veterans: PTSD and no disorder comparisons. Neuropsychology. 2002 Jan;16(1):5-14. doi: 10.1037//0894-4105.16.1.5. PMID 11853357
- [Background] Velligan DI, Kern RS, Gold JM. Cognitive rehabilitation for schizophrenia and the putative role of motivation and expectancies. Schizophr Bull. 2006 Jul;32(3):474-85. doi: 10.1093/schbul/sbj071. Epub 2006 Apr 26. PMID 16641424
- [Background] Vita A, Deste G, De Peri L, Barlati S, Poli R, Cesana BM, Sacchetti E. Predictors of cognitive and functional improvement and normalization after cognitive remediation in patients with schizophrenia. Schizophr Res. 2013 Oct;150(1):51-7. doi: 10.1016/j.schres.2013.08.011. Epub 2013 Aug 30. PMID 23998953
- [Background] Watkins LE, Sprang KR, Rothbaum BO. Treating PTSD: A Review of Evidence-Based Psychotherapy Interventions. Front Behav Neurosci. 2018 Nov 2;12:258. doi: 10.3389/fnbeh.2018.00258. eCollection 2018. PMID 30450043
- [Background] Westphal M, Olfson M, Gameroff MJ, Wickramaratne P, Pilowsky DJ, Neugebauer R, Lantigua R, Shea S, Neria Y. Functional impairment in adults with past posttraumatic stress disorder: findings from primary care. Depress Anxiety. 2011 Aug;28(8):686-95. doi: 10.1002/da.20842. Epub 2011 Jun 16. PMID 21681868
- [Background] Wetherell, J. L., & Areán, P. A. (1997). Psychometric evaluation of the Beck Anxiety Inventory with older medical patients. Psychological Assessment, 9(2), 136-144. https://doi.org/10.1037/1040-3590.9.2.136
- [Background] Wild J, Gur RC. Verbal memory and treatment response in post-traumatic stress disorder. Br J Psychiatry. 2008 Sep;193(3):254-5. doi: 10.1192/bjp.bp.107.045922. PMID 18757989
- [Background] Wild J, Warnock-Parkes E, Grey N, Stott R, Wiedemann M, Canvin L, Rankin H, Shepherd E, Forkert A, Clark DM, Ehlers A. Internet-delivered cognitive therapy for PTSD: a development pilot series. Eur J Psychotraumatol. 2016 Nov 8;7:31019. doi: 10.3402/ejpt.v7.31019. eCollection 2016. PMID 27837579
- [Background] Wills, T. A., & Fegan, M. F. (2001). Social networks and social support. In A. Baum, T. A. Revenson, & J. E. Singer(Eds.), Handbook of health psychology (pp. 209-234).Mahwah, NJ: Erlbaum.
- [Background] Wills, T. A., & Shinar, O. (2000). Measuring perceived and received social support. In S. Cohen, L. G. Underwood, & B. H. Gottlieb (Eds.), Social support measurement and intervention: A guide for health and social scientists (pp. 86-135). Oxford University Press.https://doi.org/10.1093/med:psych/9780195126709.003.0004
- [Background] Wright BK, Kelsall HL, Sim MR, Clarke DM, Creamer MC. Support mechanisms and vulnerabilities in relation to PTSD in veterans of the Gulf War, Iraq War, and Afghanistan deployments: a systematic review. J Trauma Stress. 2013 Jun;26(3):310-8. doi: 10.1002/jts.21809. Epub 2013 May 13. PMID 23670878
- [Background] Woon FL, Farrer TJ, Braman CR, Mabey JK, Hedges DW. A meta-analysis of the relationship between symptom severity of Posttraumatic Stress Disorder and executive function. Cogn Neuropsychiatry. 2017 Jan;22(1):1-16. doi: 10.1080/13546805.2016.1255603. Epub 2016 Nov 22. PMID 27875926
- [Background] Wrocklage KM, Schweinsburg BC, Krystal JH, Trejo M, Roy A, Weisser V, Moore TM, Southwick SM, Scott JC. Neuropsychological Functioning in Veterans with Posttraumatic Stress Disorder: Associations with Performance Validity, Comorbidities, and Functional Outcomes. J Int Neuropsychol Soc. 2016 Apr;22(4):399-411. doi: 10.1017/S1355617716000059. Epub 2016 Feb 19. PMID 26892753
- [Background] Wu J, Ge Y, Shi Z, Duan X, Wang L, Sun X, Zhang K. Response inhibition in adolescent earthquake survivors with and without posttraumatic stress disorder: a combined behavioral and ERP study. Neurosci Lett. 2010 Dec 17;486(3):117-21. doi: 10.1016/j.neulet.2010.07.040. Epub 2010 Jul 22. PMID 20655367
- [Background] Wykes T, Reeder C, Landau S, Matthiasson P, Haworth E, Hutchinson C. Does age matter? Effects of cognitive rehabilitation across the age span. Schizophr Res. 2009 Sep;113(2-3):252-8. doi: 10.1016/j.schres.2009.05.025. Epub 2009 Jun 12. PMID 19524409
- [Background] Xue C, Ge Y, Tang B, Liu Y, Kang P, Wang M, Zhang L. A meta-analysis of risk factors for combat-related PTSD among military personnel and veterans. PLoS One. 2015 Mar 20;10(3):e0120270. doi: 10.1371/journal.pone.0120270. eCollection 2015. PMID 25793582
- [Background] Yehuda R, Golier JA, Halligan SL, Harvey PD. Learning and memory in Holocaust survivors with posttraumatic stress disorder. Biol Psychiatry. 2004 Feb 1;55(3):291-5. doi: 10.1016/s0006-3223(03)00641-3. PMID 14744471
- [Background] Yehuda R, Golier JA, Tischler L, Stavitsky K, Harvey PD. Learning and memory in aging combat veterans with PTSD. J Clin Exp Neuropsychol. 2005 May;27(4):504-15. doi: 10.1080/138033990520223. PMID 15962694
- [Background] Yehuda R, Tischler L, Golier JA, Grossman R, Brand SR, Kaufman S, Harvey PD. Longitudinal assessment of cognitive performance in Holocaust survivors with and without PTSD. Biol Psychiatry. 2006 Oct 1;60(7):714-21. doi: 10.1016/j.biopsych.2006.03.069. PMID 17008144